CLINICAL TRIAL: NCT07370558
Title: EVIDENCE-BASED NURSING CARE AT THE BOTTOM OF THE HIERARCHY: PRACTICE, BARRIERS, AND FACILITATORS
Brief Title: EVIDENCE-BASED NURSING CARE AMONG SURGICAL NURSES
Status: Not yet recruiting | Type: Observational
Sponsor: AKİF BULUT (Other)
Responsible Party: Sponsor-Investigator, AKİF BULUT, Assistant Investigator, Uludag University
Organization: Uludag University (Other)
Other Study IDs: 2025-9/6
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Nurse's Role

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical nurses: Nurses working in surgical clinics and operating rooms
  Interventions: Other: Measuring evidence-based nursing knowledge and practice levels using a scale

INTERVENTIONS:
Other: Measuring evidence-based nursing knowledge and practice levels using a scale — Turkish Ministry of Health Uludağ University Faculty of Medicine Hospital Nurses working in surgical clinics will be assessed using the Research Use Barriers Scale and the Evidence-Based Practice Usage Scale to determine their levels of evidence-based nursing practice, the barriers they encounter, and the facilitating factors.

SUMMARY:
Background: There is a limited number of studies in Turkey that jointly evaluate the evidence-based practice levels of nurses working in surgical units, the barriers they encounter in practice, and the facilitating factors that support practice. In particular, understanding the extent to which evidence-based nursing practice beliefs predict evidence-based care practice behaviors is important for designing in-house training programs, creating clinical guidelines, and developing in-service mentoring systems.

Purpose: This research was conducted to reveal the levels of evidence-based nursing practice among nurses working in surgical units, identify barriers to implementation, and define factors that facilitate implementation. It is anticipated that the findings will guide clinical managers, education planners, and policy developers in creating evidence-based improvement strategies.

Methodology: The research is a descriptive-cross-sectional study. The population consists of nurses working in the Surgical Clinics at Uludağ University Faculty of Medicine Hospital in Bursa, Turkey (N:350). The sample calculation for the study was performed using the known population sample method. The minimum number of individuals required in the sample was calculated using the Raosoft sample calculation tool, yielding a sample size (n) of 184 when a 5% margin of error and a 95% confidence interval were applied.

ELIGIBILITY:
Inclusion Criteria:

* Working as a Clinical Nurse (in surgical areas) at Uludağ University Faculty of Medicine Hospital, Ministry of Health, Republic of Turkey,
* Agreeing to participate in the study as a volunteer,
* Not having any visual, auditory, or psychological problems that would prevent them from completing the questionnaire and scales,
* Being a graduate of nursing school.

Exclusion Criteria:

* Not working as a nurse in the Clinical Department (surgical fields) at Uludağ University Faculty of Medicine Hospital, Ministry of Health of the Republic of Turkey,
* Not agreeing to participate in the research as a volunteer,
* Having any visual, auditory, or psychological problems that would prevent them from completing the questionnaire and scales,
* Not being a graduate of nursing school.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses working in the Clinical Department (Surgical fields) at Uludağ University Faculty of Medicine Hospital, Ministry of Health of the Republic of Turkey
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Evidence-Based Practice Usage Scale | 6 months
  It includes 18 items, including creating a PICO (Population, Intervention, Comparison, Outcome) question about the applications, using evidence to change clinical practices, and sharing the collected data results with colleagues. A five-point frequency scale (ranging from 0 = '0 times' to 4 = '>8 times') is used to indicate how often participants performed each item in the last eight weeks, with a total score ranging from 0 to 72. A higher score indicates greater use of evidence-based nursing care.

SECONDARY OUTCOMES:
Research Usage Barriers Scale | 6 months
  The scale consists of four subdimensions: nursing, practice, research, and presentation. The "Nursing" subdimension contains eight items that assess nurses' value, skills, and awareness of research, while the "Practice" subdimension contains eight items that assess perceived barriers and limitations in the work environment. The "Research" sub-dimension consists of 6 items that assess the quality of research, while the "Presentation" sub-dimension consists of 6 items that assess comprehensibility and usability. A score of 1 on the four-point Likert scale means "no obstacle," 2 means "minor obstacle," 3 means "moderate obstacle," and 4 means "major obstacle." Alternatively, the option "0-no opinion" is also included in the scale, but these responses are not included in the scoring. Therefore, the overall average score of the scale ranges from 30 to 120 points.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Eda Tekin, Assit. Prof., Principal Investigator — Mudanya University

IPD SHARING:
Plan to Share IPD: No